CLINICAL TRIAL: NCT06155656
Title: Acute Effects of Pea Proteins With Different Degrees of Processing on Postprandial Metabolism in Healthy Women and Men
Brief Title: Effects of Pea Proteins With Different Degrees of Processing on Postprandial Metabolism in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); University of Bonn, Department of Nutrition and Food Sciences, Food Sciences (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Sarah Egert, Prof PhD, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AlProPlant-HS1
Record Dates: First submitted 2023-11-07; First posted 2023-12-04 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Plasma Amino Acid Appearance and Disappearance; Postprandial Metabolic Events
Keywords: Postprandial metabolic events
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pea concentrate (Experimental): Participants randomized to receive a soup containing 25 g of protein from pea protein concentrate
  Interventions: Other: Pea protein concentrate
- Pea isolate (Experimental): Participants randomized to receive a soup containing 25 g of protein from pea protein isolate
  Interventions: Other: Pea protein isolate
- Pea extrudate (Experimental): Participants randomized to receive a soup containing 25 g of protein from pea protein extrudate
  Interventions: Other: Pea protein extrudate
- Whey (Active Comparator): Participants randomized to receive a soup containing 25 g of protein from whey protein
  Interventions: Other: Whey protein

INTERVENTIONS:
Other: Pea protein concentrate — Ingestion of a soup containing 25 g of protein from pea protein concentrate
  Arms: Pea concentrate
Other: Pea protein isolate — Ingestion of a soup containing 25 g of protein from pea protein isolate
  Arms: Pea isolate
Other: Pea protein extrudate — Ingestion of a soup containing 25 g of protein from pea protein extrudate
  Arms: Pea extrudate
Other: Whey protein — Ingestion of a soup containing 25 g of protein from whey protein
  Arms: Whey

SUMMARY:
The aim of this study is to investigate the postprandial metabolic responses to plant-based protein ingredients of different degrees of processing (pea protein concentrate, isolate, and extrudate) and in comparison to whey protein in healthy adults. Therefore, young healthy subjects consume 4 test meals with 25 g of protein from pea protein concentrate, pea protein isolate, pea protein extrudate or whey protein in a randomized order. In a postprandial period of 6 hours, parameters of protein and glucose metabolism (i.a. plasma amino acids), gastric emptying and hunger/satiety are analysed. It is assumed that the plasma amino acid profile after plant protein ingestion differs depending on processing level of the protein ingredients and in comparison to whey protein.

DETAILED DESCRIPTION:
In a randomized crossover-design, 20 healthy women and men consume 4 test meals containing either 25 g of protein from plant protein ingredients (pea protein concentrate, isolate, or extrudate) or whey protein together with 1 g paracetamol, which is used as a marker for gastric emptying.

During a postprandial period of 6 hours parameters of protein metabolism (e.g. amino acids in plasma and urine), glucose metabolism (plasma glucose, serum insulin) and gastric emptying rate (based on plasma paracetamol) are analysed. Furthermore, subjective hunger/satiety and acceptance of the meals are assed using visual analogue scales. Each intervention arm will be separated by a washout period of at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* metabolically healthy
* normal weight (BMI: 18,5 - 24,9 kg/m2)
* written informed consent

Exclusion Criteria:

* pregnancy, lactation
* hypo- or hypertension
* underweight or overweight/obesity
* food intolerances and allergies (especially milk protein, pea, celery)
* malabsorption syndromes
* gastrointestinal diseases
* thyroid diseases
* diabetes mellitus type 1 and type 2
* impaired kidney or liver function
* anaemia
* blood coagulation disorders
* irregular menstrual cycle
* endometriosis, severe menstrual problems
* hormonal contraception
* regular use of medications (especially habitual use of paracetamol or medications that may interact with paracetamol)
* hypersensitivity to paracetamol
* body weight below 50 kg
* alcohol abuse
* glucose-6-phosphate dehydrogenase deficiency
* Gilbert's syndrome
* vegan diet
* eating disorders (especially anorexia nervosa, bulimia nervosa)
* smoking
* participation in another study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Amino acid profile in blood | Postprandial period of 5 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 300 minutes)
  Analysis of amino acid profile in plasma (nmol/ml)

SECONDARY OUTCOMES:
Parameters of protein metabolism in blood I | Postprandial period of 5 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 300 minutes)
  Analysis of urea (mg/dL and mol/L) in blood
Parameters of protein metabolism in blood II | Postprandial period of 5 hours (Time points: fasting (0) and 60, 120, 180, 240 and 300 minutes)
  Analysis of nitrogen (mg/dL) in blood
Parameters of glucose metabolism in blood I | Postprandial period of 5 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 300 minutes)
  Analysis of glucose (mg/dL and mmol/L) in blood
Parameters of glucose metabolism in blood II | Postprandial period of 5 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 300 minutes)
  Analysis of insulin (nmol/L and pmol/L) in blood
Gastric emptying rate | Postprandial period of 5 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 300 minutes)
  Analysis of gastric emptying rate based on paracetamol kinetics in blood (µg/mL)
Hunger/satiety and acceptance of the meals | Postprandial period of 5 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 300 minutes)
  Assessment of subjective hunger/satiety and acceptance of the meals by validated visual analogue scale questionnaires (e.g., 0 = not hungry at all, 10 = very hungry)
Uric acid in blood | Postprandial period of 5 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 300 minutes)
  Analysis of uric acid (mg/dL and mmol/L) in blood
Copper in blood | Postprandial period of 5 hours fasting (0) and 60, 120, 180, 240 and 300 minutes)
  Analysis of copper (µg/l) in blood
Zinc in blood | Postprandial period of 5 hours fasting (0) and 60, 120, 180, 240 and 300 minutes)
  Analysis of zinc (µg/l) in blood
Iron in blood | Postprandial period of 5 hours fasting (0) and 60, 120, 180, 240 and 300 minutes)
  Analysis of iron (µg/l) in blood
Selenium in blood | Postprandial period of 5 hours fasting (0) and 60, 120, 180, 240 and 300 minutes)
  Analysis of selenium (µg/l) in blood
Amino acid profile in urine | Postprandial period of 5 hours
  Analysis of amino acids in urine (nmol/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Egert, Prof PhD, Principal Investigator — Germany University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No